CLINICAL TRIAL: NCT04751500
Title: The HYsteroscopic Miscarriage MaNagement (HYMMN) Trial
Brief Title: The HYsteroscopic Miscarriage MaNagement Trial: A Pilot RCT Investigating a Novel Management Pathway for RPOC
Acronym: HYMMN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham Women's and Children's NHS Foundation Trust (Other)
Collaborators: Tommy's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 276909; 20/WM/0287 (Other: HRA and Health and Care Research Wales (HRCW))
Record Dates: First submitted 2021-01-29; First posted 2021-02-12 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Retained Products After Miscarriage
Keywords: ultrasound; hysteroscopy; miscarriage; retained products of conception
MeSH Terms: conditions — Abortion, Incomplete; Abortion, Spontaneous | interventions — Watchful Waiting; Practice Management, Medical; Misoprostol; Mifepristone; Anti-Bacterial Agents; Amoxicillin-Potassium Clavulanate Combination; Metronidazole; Clindamycin; Dilatation

STUDY DESIGN:
Intervention Model Description: The study involves two phases: 1) All recruited women will be scanned for RPOC at 8 weeks post-miscarriage diagnosis. 2) Women that have RPOC on this scan will then be randomised in a 1:1 manner to either outpatient hysteroscopy or standard treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient Hysteroscopy (Experimental): Outpatient hysteroscopic morcellation of retained products of conception
  Interventions: Procedure: Outpatient hysteroscopy
- Standard Treatment (Active Comparator): Standard treatment of retained products of conception in the form of expectant management, medical management, antibiotic therapy and/or surgical management (manual vacuum aspiration/suction curettage/dilatation and curettage)
  Interventions: Behavioral: Expectant management; Drug: Medical management; Drug: Antibiotic; Procedure: Surgical management

INTERVENTIONS:
Procedure: Outpatient hysteroscopy — Direct visualisation and careful extraction of retained pregnancy tissue using a specific hysteroscopic technology known as a hysteroscopic tissue retrieval system.
  Arms: Outpatient Hysteroscopy
Behavioral: Expectant management — Leaving the retained pregnancy tissue alone to pass by itself
  Arms: Standard Treatment
Drug: Medical management — Giving medications to contract the womb to pass the retained pregnancy tissue
  Other Names: misoprostol; mifepristone
  Arms: Standard Treatment
Drug: Antibiotic — Giving antibiotics to reduce any inflammation/infection caused by the retained pregnancy tissue allowing it to pass by itself
  Other Names: Augmentin; Co-amoxiclav; Metronidazole; Clindamycin
  Arms: Standard Treatment
Procedure: Surgical management — Passing a small cannula/catheter/currette into the womb and mechanically scraping the womb lining to remove the retained pregnancy tissue
  Other Names: manual vacuum aspiration; suction evacuation of the uterus; dilatation and currettage
  Arms: Standard Treatment

SUMMARY:
Pregnancy tissue can be found remaining in the womb in up to 20% of women following a miscarriage. These "retained products of conception" (RPOC), which are diagnosed by transvaginal ultrasound, can cause prolonged bleeding, pain, infection, impaired fertility and therefore further psychological distress. Ineffective medical and surgical interventions place considerable burden on affected women and utilise scarce health care resources. Additionally, surgery is performed 'blindly' using a suction tube or metal curette where risks include perforation of the womb and scarring of the womb lining, both of which lead to delayed fertility and in the worst circumstances, infertility.

There is no current guidance on how to best investigate and manage RPOC. New surgical equipment allows RPOC removal under vision, using a specially designed telescope placed inside the womb (hysteroscopy). This precise technique may more successfully and less traumatically remove RPOC, minimising ongoing bleeding, the risk of womb perforation and scar tissue formation, thereby reducing the risk of infertility.

The investigators propose a pilot randomised controlled trial using routine transvaginal ultrasound to diagnose RPOC in women who choose non-surgical management of a first-trimester (≤14 weeks) miscarriage. This scan will be done 8 weeks post-miscarriage diagnosis. Women who have RPOC on this scan will be randomised (in a 1:1 ratio) to receive outpatient hysteroscopy ('OPH') or 'standard treatment' (expectant, medical, surgical and/or antibiotic treatment).

Women who had RPOC will be followed-up at 14 weeks after randomisation to explore clinical outcomes (symptoms, quality of life) and use of additional healthcare resources (e.g. additional investigations / treatments / hospitalisations). All patients, no matter whether they were diagnosed with RPOC or not, will be followed up at 26 weeks and 52 weeks after randomisation/ultrasound scan to determine clinical pregnancy rates and pregnancy outcomes. All patients who have had a miscarriage or have not fallen pregnant since entering the trial will be offered a hysteroscopy to see if there are any conditions affecting the womb lining which may be contributing to pregnancy failure.

DETAILED DESCRIPTION:
The diagnosis of retained products of conception (RPOC) following miscarriage causes physiological and emotional stress to women and their partners. Additional hospital visits, inpatient admissions and non-evidence-based treatments impose an additional burden on women and healthcare services. Ineffective medical and surgical treatments can prolong symptoms such as bleeding, pain and psychological distress which impacts adversely on quality of life. In addition, future fertility can be delayed or worse, permanently impaired, because of damage and scarring of the womb lining arising from chronic infection or mechanical trauma after conventional 'blind' mechanical evacuation of the uterine cavity.

Recent technological advances in hysteroscopy allow RPOC to be directly visualised and simultaneously removed with greater precision and less trauma to the endometrium with promising results. These 'hysteroscopic tissue removal systems' represent the latest advance in uterine surgery. This technology allows complete excision and removal of intrauterine pathology under direct vision, including removal of RPOC in the inpatient and more recently, the outpatient setting with complete resection and resolution of symptoms without apparent complications. Current evidence suggests that hysteroscopic resection of RPOC is associated with the formation of less intrauterine adhesions, lower rates of incomplete evacuation, and shorter time to subsequent conception, but is based on limited numbers of studies, too small sample sizes to statistically detect differences between treatments, poor reporting of confounders and the absence of randomised studies.

To date, there are no randomised controlled trials investigating the use of outpatient hysteroscopy in the management of RPOC against standard treatment. The investigators therefore aim to perform a pilot randomised control trial to assess the feasibility of undertaking a future substantive full-scale trial to compare routine transvaginal ultrasound scanning and outpatient hysteroscopy for the treatment of RPOC against current standard practice to see if it is more effective in improving fertility and minimising symptomatic morbidity. Furthermore, health service resource use will be evaluated against clinical outcomes to determine the cost-effectiveness of this new pathway.

All women who choose non-surgical management of a first trimester (≤14 weeks gestation) miscarriage will be eligible for recruitment into the study, where informed consent will be taken and baseline assessments will be conducted.

All patients who then have RPOC diagnosed on transvaginal ultrasound scan (TVS) at 8 weeks after the diagnosis of their miscarriage will then be randomised (in a 1:1 ratio) to receive outpatient hysteroscopy ('OPH') or 'standard treatment'. At 'OPH', if RPOC are present, then these will be removed on an intention-to-treat basis. If randomised to the 'standard treatment' arm, management will be based according to current practice (expectant, medical, antibiotic, surgical treatment). Immediately after OPH, all women will be asked to complete a questionnaire exploring the acceptability of the procedure and clinicians will be asked to complete a questionnaire exploring the efficacy of OPH in diagnosing and removing RPOC.

For those who had RPOC, regardless of which treatment they were randomised to, face-to-face consultations will be performed at 14 weeks post-randomisation. These will explore clinical outcomes (symptoms and generic quality of life) and use of additional healthcare resources (e.g. additional investigations / treatments / hospitalisations). All patients, no matter whether they were diagnosed with RPOC or not, will be followed up at 26 weeks and 52 weeks post-randomisation to determine clinical pregnancy rates and pregnancy outcomes. All patients who have had a miscarriage or have not fallen pregnant since entering the trial will be offered the chance to undergo a hysteroscopy to see if there is any scar tissue, chronic RPOC or other conditions affecting the womb lining which may be contributing to pregnancy failure; this data will be collected. At this point, patients will discharged from the trial.

The sample size of a future substantive study will partly be determined by the results of this study. This study will aim to recruit 200 women to give a better idea of the number of women with RPOC and the numbers willing to be recruited. After recruitment, the investigators will aim to scan 200 women over a six-month period. Predicated upon a sonographic RPOC rate of 20%, 40 women are expected to have RPOC; 20 women would be randomised to 'OPH' and 20 women to 'nOPH'.

ELIGIBILITY:
Inclusion Criteria:

* Women above 18 years
* Women choosing either expectant or medical management of a first-trimester miscarriage ≤14 weeks gestation
* Women wanting to conceive as soon as possible after their miscarriage
* Consent to trial processes: (1) undergo follow-up with transvaginal ultrasound for the investigation of RPOC; (2) be randomised to outpatient hysteroscopy for confirmation and treatment or standard management; (3) accept trial follow up procedures - questionnaires, telephone interviews

Exclusion Criteria:

* Women below 18 years
* Women with findings suspicious of gestational trophoblastic disease
* Women with fever (≥38°C) or sepsis secondary to genital tract infection/endometritis
* Women who are unable to understand spoken and written English

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Number of eligible patients | During recruitment - 6 months
  The number of patients approached that fulfill the eligibility criteria for entry into the trial
Proportion of patients enrolled into the trial | During recruitment - 6 months
  The proportion of eligible women that agree to participate in the trial
Proportion of patients attending scan | At ultrasound scan 8 weeks post-miscarriage diagnosis
  The proportion of women that attended the hospital for their 8-week post-miscarriage ultrasound scan
Proportion of patients attending outpatient hysteroscopy (if randomised to this treatment) | During outpatient hysteroscopy (if randomised to this treatment)
  Of the women randomised to hysteroscopic treatment of RPOC, the proportion that attended their appointment
Proportion of patients attending 14-week follow-up | 14-week follow up
  The proportion of women that attended follow-up at 14 weeks
Proportion of patients attending 26-week follow-up | 26-week follow up
  The proportion of women that attended follow-up at 26 weeks
Proportion of patients attending 52-week follow-up | 52-week follow up
  The proportion of women that attended follow-up at 52 weeks
Acceptability of trial to eligible women | Up to 8 months
  To determine why patients decline participation into the trial or withdraw after consent
Acceptability of ultrasound scan to patients | At ultrasound scan 8 weeks post-miscarriage diagnosis
  Acceptability of ultrasound scan to patients as recorded on a questionnaire given to the woman after their ultrasound scan on a 5-point Likert scale
Acceptability of outpatient hysteroscopy to patients | During outpatient hysteroscopy (if randomised to this treatment)
  Acceptability of outpatient hysteroscopy to patients, if randomised to this treatment, as recorded on a questionnaire given to the woman after their hysteroscopy on a 5-point Likert scale
Robustness of data collection tools | From recruitment of first patient to end of trial (up to 20 months)
  Assessing the completion of the patient and clinician questionnaires during the course of the study to determine how robust/appropriate the data collection tools are (we would expect at least 90% of the forms to be filled out)

SECONDARY OUTCOMES:
Clinical pregnancy rates | Assessed at 26 and 52 weeks post-randomisation/ultrasound scan
  Clinical pregnancy rates
Time to next pregnancy | Assessed at 26 and 52 weeks post-randomisation/ultrasound scan
  Time to next pregnancy
Symptoms | 14 weeks post-randomisation/ultrasound scan
  Number of patients with menstrual bleeding, abdominal pain and vaginal discharge symptoms
Impact on quality of life | 14 weeks post-randomisation/ultrasound scan
  Adapted EuroQol- 5 Dimension (EQ-5D-5L)
Impact on work | 14 weeks post-randomisation/ultrasound scan
  Time absent from work
Healthcare resource use | 14 weeks post-randomisation/ultrasound scan
  Number of consultations, scans, inpatient hospital admissions, overnight stays, treatments administered
Patient satisfaction | 14 weeks post-randomisation/ultrasound scan
  Patient satisfaction of trial process (i.e. ultrasound scan +/- treatment for retained products of conception) on a 10cm visual analogue scale
Procedural findings at ultrasound | During ultrasound scan 8 weeks post-miscarriage diagnosis
  Ultrasound findings of patients categorised into whether RPOC are present or not. If RPOC are present, dimensions of RPOC (in millimeters) and presence of vascularity (yes/no) are to be recorded.
Ease of diagnosis of retained products of conception (RPOC) | During ultrasound scan 8 weeks post-miscarriage diagnosis
  Ease of diagnosis of retained products of conception on ultrasound scan by scan operator on a 10cm visual analogue score
Procedural findings at outpatient hysteroscopy (in women randomised to this treatment) | During outpatient hysteroscopy (in women randomised to this treatment)
  Hysteroscopic findings/procedural success in women randomised to outpatient hysteroscopy
Ease of removal of RPOC during outpatient hysteroscopy (in women randomised to this treatment) | During outpatient hysteroscopy (in women randomised to this treatment)
  Ease of hysteroscopic morcellation of RPOC and procedural success from clinician perspective, recorded on a 10cm visual analogue scale
Pain experienced by patients undergoing outpatient hysteroscopy (in women randomised to this treatment) | During outpatient hysteroscopy (in women randomised to this treatment)
  Pain experienced by patients undergoing outpatient hysteroscopy on a 10cm visual analogue scale
Proportion of women with adverse pregnancy outcomes at 52 weeks | 52 weeks post-randomisation/ultrasound scan
  Proportion of women with no pregnancy or failed pregnancy (ectopic pregnancy, miscarriage) at 52-week follow up
Hysteroscopic findings in women with adverse pregnancy outcomes at 52 weeks | During outpatient hysteroscopy after 52 weeks post-randomisation/ultrasound scan
  Hysteroscopic findings in women with adverse pregnancy outcomes at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: T Justin Clark, FRCOG, Principal Investigator — Birmingham Women's NHS Foundation Trust
Locations (1):
- Birmingham Women's Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Any physical paperwork containing identifiable data will be kept in an access-controlled, secured room inside the Birmingham Women's and Children's NHS Foundation Trust in a secure locked office. Anonymised data will be uploaded from the site office to the electronic Remote Data Capture system (eRDC) system, hosted on the University of Birmingham server. The security of the System is governed by the policies of the University of Birmingham. The University's Data Protection Policy and the Conditions of Use of Computing and Network Facilities set out the security arrangements under which sensitive data should be processed and stored. The Study Centre has arrangements in place for the secure storage and processing of the study data which comply with the University of Birmingham policies.